

## **Analysis Strategy**

We conducted all analysis in IBM SPSS V19. We used the Generalized Linear Model to examine the between-condition change over time on study outcomes. The effects of primary interest were those reflecting the effects of WILLOW. For outcomes measured at baseline and follow-up points, that was the Time X Condition effects (measuring between-condition change from baseline). For outcomes measured only at follow-up points (e.g., therapeutic alliance and use of evidence-based therapy tasks), that was the Condition effects since they would represent average between-condition differences during the time patients received services. As previously mentioned, providers completed questionnaires for each study patient they treated. Hence, the provider sample size reflects the number of patients they answered about, not the number of providers. Several providers participated in the study concurrently with multiple patients. Patients were included in the analyses only if they attended five or more sessions with a participant provider.

Preliminary analyses provided important information guiding our strategy. First, we found no statistically significant differences between conditions on baseline measures. Second, we computed the design effects due to this nested design to determine the extent to which the intraclass correlation due to clustering and size of the cluster affected the analyses. Design effects ranged up to 1.8. Because all were under 2.0, we did not adjust analyses to account for clustering effects (Muthén & Satorra, 1995). For providers meeting participating in both studies, we used their Study 1 data for outcomes except for outcomes measured only in Study 2. For those outcomes, we used their Study 2 data.

## References

Muthén, B.O. & Satorra, A. (1995). Complex sample data in structural equation modeling. *Sociological Methodology*, *25*, 267-316. doi: 10.2307/271070